CLINICAL TRIAL: NCT03499665
Title: Assessment The Effects of Proprioceptive Neuromuscular Facilitation, Myofascial Releasing Maneuvers and Home Exercises on Pain and Jaw Function in Patients With Bruxism
Brief Title: The Effects of Proprioceptive Neuromuscular Facilitation, Myofascial Releasing Maneuvers and Home Exercises on Pain and Jaw Function in Patients With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Elisa Çalışgan, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/98
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Exercise; Bruxism; Myofascial
Keywords: Bruxism; Pain; Exercises; Myofascial; Releasing
MeSH Terms: conditions — Motor Activity; Bruxism; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, Randomized Controlled Study
Who Masked: Participant
Masking Description: Participants didn't know taking which exercise treatment methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNF, Myofascial Releasing Maneuvers, Home Exercise Group (Experimental): This group of patients received patients with bruxism. It was applied proprioceptive neuromuscular facilitation (PNF), myofascial releasing maneuvers and home exercises.
  Interventions: Behavioral: PNF, Myofascial Releasing Maneuvers, Home Exercise Group
- Myofascial Releasing Maneuvers and Home Exercises Group (Active Comparator): This group of patients received patient with bruxism. It was applied myofascial releasing maneuvers and home exercises.
  Interventions: Behavioral: Myofascial Releasing Maneuvers and Home Exercises Group
- Control Group (Active Comparator): This group of patients received patient with bruxism. It was applied conventional treatment and no myofascial releasing or Proprioceptive Neuromuscular Facilitation exercises were applied.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: PNF, Myofascial Releasing Maneuvers, Home Exercise Group — For Group 1 (n:20), the PNF, myofascial releasing and home exercises were used to decrease pain, jaw restriction and improve functional mobility on the masseter, lateral and medial pterygoid, buccinator, temporalis, orbicularis oris, orbicularis oculi, upper side of trapezius muscle, splenius, scalenous, and cervical extensor muscle in 20 patients with bruxism, for 2 and 6 weeks after pre-evaluation. PNF, myofascial releasing and home exercises were administered for 2 weeks, followed by 3 sets of 10 repeat home exercises and 6 weeks under physiotherapist control.
  Arms: PNF, Myofascial Releasing Maneuvers, Home Exercise Group
Behavioral: Myofascial Releasing Maneuvers and Home Exercises Group — In Group 2 (n:15), as myofascial releasing and home exercise group,final evaluation was made with 10 sets of myofascial releasing and home exercises for 2 and 6 weeks.
  Arms: Myofascial Releasing Maneuvers and Home Exercises Group
Behavioral: Control Group — In Group 3 (n:17), as the control group, no myofascial releasing or Proprioceptive Neuromuscular Facilitation exercises were applied.
  Arms: Control Group

SUMMARY:
This study was planned to evaluate the effects of proprioceptive neuromuscular facilitation, myofascial releasing maneuvers and home exercises on pain and jaw function in patients with bruxism aged 16-50 years .

DETAILED DESCRIPTION:
Bruxism is different from temporomandibular joint disease because of long periods of muscle contraction. It is considered an eloquent contributory factor in the etiology of temporomandibular disorders (TMD). The incidence of bruxism is estimated to be approximately between 5% and 10% of the adult population. Especially long term contraction of masseter, temporalis and medial pterygoid muscle cause restriction of opening mouth, problem of closing the jaw, problems of chewing, articulation, movement of tongue. Bruxism is common illness which is seen with in mood disorders such as anxiety and depression. According to Orofacial Pain Guidelines, Bruxism is a diurnal or nocturnal parafunctional activity including clenching, bracing, grinding and gnashing of the teeth. An oral habit consisting of involuntary rhythmic or spasmodic nonfunctional horizontally and vertically gnashing, grinding or clenching of teeth, in other than chewing movements of the mandible, this may bring about occlusal trauma.

The factors involving anatomical- morphological, psychophysiological, pathophysiological factors and other cause diurnal or nocturnal bruxism. Researchers say that genetics account for 30 to 50 percent of bruxism with nocturnal or diurnal and behaviour, environmental account for the remainder. Dental malocclusion, anatomical- morphological differences, anomalies of the oro-facial region (condyles height asymmetry, hypognathism, larger cranial, bizygomatic width, rectangular form of dental arch of maxilla, rectangular morphology of face) psychophysiological reasons including stress in which result from emotional, physical, psychosocial stimulation, anxiety, depression, psychosomatic disorders, personality disorders such as hyperactivity, hysteria, aggressiveness, tendency of perfectionist affect oral function and cause bruxism . Sleep disturbances known as especially sleep apnea, behaviour disorder during REM ( rapid eye movement) and Non-REM (non- rapid eye movement) sleep stimulate of nocturnal bruxism. Consume of drug such as antidepressants (SSRI) have suppression and stimulate effects on patients seen. Vulnerable disorders of central dopaminergic neurotransmission, hemifacial spasm, stroke brain haemorrhage, Huntington chorea, Parkinson disease give rise to bruxism. While the acute use of L- dopa drugs inhibits bruxism activity, the chronic use of L- dopa in patients with Parkinson lead to bruxism. This situation is same effect with antiepileptic drugs. According to some criteria bruxism may be categorized by when it appears awake bruxism which is presented when the person is awake, sleep bruxism which is presented when the person is sleep and combined bruxism which is presented when seen two situations . By etiology researcher classified with primary or idiopathic bruxism which no apparent cause is known. Secondary bruxism occurs with diseases (coma, ictus, cerebral palsy), medicinal products (e.g. antipsychotic medication), drugs (such as amphetamines, ecstasy). Bruxism classified motor activity type of tonic, phasic, combined and by current or past presence such as past bruxism, current or present bruxism. Sleep bruxism major seen during REM and Non- REM sleep and is the most common type of bruxism than others. Its incidence has been the highest in childhood (vitally 14%) and decreases from about 8% in younger adults to almost 3% in elderly people called negative correlation . In awake bruxism is an involuntary activity of the jaw muscles that is characterized, by jaw clenching, by tooth gnashing and/or grinding. During sleep bruxism, both clenching and tooth grinding are observed. Sleep bruxism can lead to tooth destruction, temporomandibular pain and crepitation, headaches and grinding sounds . A lot of patients are complain of jaw tightness and grinding sounds daily or nightly, while others said these infrequently. In cases of severe and frequent sleep bruxism, the variation of the number of episodes per hour of sleep is 25%, and the variation of tooth-grinding frequency is 53.5%. Symptoms of bruxism are abnormal tooth wear, teeth gliding or clenching, sounds because of clenching and gliding, gingival inflammation, headache, ocular pain, limited opening of mouth, decrease of salivary flow, erythema, photosensitivity, tinnitus, ear plugging sensation, temporomandibular pain (TMP), destruction and click sounds. When overtime in patients have chronic bruxism will bring about hypertrophy of masseter and temporal muscles. Therefore, patients facial appearance seems either too square or too masculine. One of the general symptoms are jaw clicking, when opening of mouth; oral muscle deviation to one side, pain in cheek muscles, uncontrollable movement of jaw. Effects of bruxism on throat are swallowing difficulties, voice irregularities, frequence coughing, feeling of foreign things in throat. In addition it causes neck problems such as pain of the shoulders and ache of back, lack of mobility, stiffness, pain of neck. Facial changing are seen patients with bruxism skin and facial muscles atrophy due to not using, vermilion thighs, dropping corners of mouth., Treatment of bruxism includes botulinum toxin, using occlusal splint, perioral rejuvenation and an antidepressant drugs. Our study shows that self-care, Proprioceptive neuromuscular facilitation exercise, myofascial thingness and home exercise including facial muscle stimulation for weight transform between bilateral side. Mainly self-care is more important than others. Therefore, we informed patients about causes, etiology, triggered effects, prevalence, incidence of bruxism, normal treatment of bruxism and our treatment stages and goals. It includes that patients are aware of bruxism. When the patients who have bruxism diagnosis, feel pain on face muscle, they need to use ice on jaw muscle. In addition they avoid eating rigid, hard stick, candy and nuts. Also, they avoid chewing gum and elastic rating, avert jaw movement forward. They should sleep the least 8 hours and need to learn stretching exercise to restore of the facial muscle and joints. In addition flexibility and stretching training of orbicularis oris and oculi, extensor muscle stabilization exercises are used for bruxism treatment. Main purpose of this study is to evaluate of the effects of proprioceptive neuromuscular facilitation , myofascial releasing maneuvers and home exercises on temporomandibular joint pain and jaw function in patients with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Having bruxism and TMJ (Temporomandibular Joint) pain,
* Bruxism patients aged 16-50 years
* At the level that can make mental evaluations,
* Will be able to adapt to the training program,
* To be involved in voluntary work,
* Individuals who have been given their informed consent

Exclusion Criteria:

Patients who are not between the ages of 16-50, who have a health problem, can not make mental evaluations, can not adapt to the education program, and refuse to participate in the study will not be included.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-02-04 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Change from pain (Visual Analog (VAS) Scale ) of patients with bruxism at 6 weeks. | 6 weeks
  The severity of pain was evaluated using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (intolerable pain).The VAS scale is recommended for evaluation because of highly reliability.

SECONDARY OUTCOMES:
Change from restriction of jaw movement (The Jaw Functional Limitation Scale ) of patients with bruxism at 6 weeks. | 6 weeks
  The Jaw Functional Limitation Scale is a scale assessing the restriction of jaw movement. It consists of 8 items related to normal daily functions of the mouth, such as chewing, yawning, swallowing and smiling, with each item scored on a scale of 0 (no restriction) to 10 (high restriction), thus total scores range from 0 -80 (8, 11).

OTHER OUTCOMES:
Change from bad oral habits(The Oral Behaviour Checklist) of patients with bruxism at 6 weeks. | 6 weeks
  The Oral Behaviour Checklist consists of 21 questions about bad oral habits. This scale is answered as a 5-point Likert scale with the responses of never, occasionally, sometimes, often, and always. The total points of the scale range from 0 to 84 .

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)